CLINICAL TRIAL: NCT07150455
Title: Evaluation of Myocardial Function by Global Longitudinal Strain (GLS) Measurement in 2D Echocardiographic Examination of Patients With Fibromyalgia
Brief Title: Evaluation of Myocardial Function by Global Longitudinal Strain (GLS) Measurement in 2D Echocardiography of Patients With Fibromyalgia
Acronym: GLS in FM
Status: Enrolling by invitation | Type: Observational
Sponsor: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Nadide Koca, Physical Medicine & Rehabilitation Specialist, Ankara Training and Research Hospital
Other Study IDs: AnkaraTRH-FTR-NK-07
Record Dates: First submitted 2025-08-25; First posted 2025-09-02 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-08

CONDITIONS: Fibromyalgia (FM); Subclinical Ventricular Dysfunction; Myocardial Function
Keywords: Fibromyalgia; Global Longitudinal Strain (GLS); 2D Echocardiography; Speckle Tracking Echocardiography; Fibromyalgia Impact Questionnaire (FIQ); Autonomic Dysfunction; Left Ventricular Function
MeSH Terms: conditions — Fibromyalgia; Primary Dysautonomias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fibromyalgia Patients: Participants aged 18-50 years diagnosed with fibromyalgia according to the 2010 American College of Rheumatology (ACR) criteria. All participants in this group will undergo 2D speckle-tracking echocardiography, including Global Longitudinal Strain (GLS) measurement, for evaluation of myocardial function. No drug or device intervention is administered.
  Interventions: Other: Echocardiographic Assessment (2D Speckle Tracking)
- Healthy Controls: Age- and sex-matched volunteers without fibromyalgia, presenting with mechanical low back pain, otherwise healthy.
  Interventions: Other: Echocardiographic Assessment (2D Speckle Tracking)

INTERVENTIONS:
Other: Echocardiographic Assessment (2D Speckle Tracking) — All participants will undergo standardized 2D echocardiographic examination including Global Longitudinal Strain (GLS) measurement. No drug or device intervention is applied.

SUMMARY:
Fibromyalgia (FM) is a chronic pain syndrome that affects multiple body systems and is often associated with fatigue, sleep disturbances, anxiety, and other comorbidities. Increasing evidence suggests that FM is also linked to cardiovascular dysfunction due to autonomic imbalance, sympathetic overactivity, and endothelial dysfunction. Patients with FM may therefore be at higher risk of developing subclinical ventricular dysfunction even before overt cardiovascular disease becomes apparent.

Traditional echocardiographic evaluation of left ventricular function is based on ejection fraction (LVEF). However, LVEF has important limitations. It may remain normal despite underlying myocardial impairment, is strongly influenced by loading conditions, and often fails to detect early myocardial dysfunction. Recent advances in echocardiography allow for the assessment of Global Longitudinal Strain (GLS), a sensitive and reproducible measure of myocardial deformation. GLS abnormalities can be detected earlier than changes in LVEF and are predictive of future declines in ejection fraction.

This study aims to evaluate myocardial function in fibromyalgia patients using GLS obtained by two-dimensional speckle-tracking echocardiography (2D-STE). By comparing FM patients with age- and sex-matched healthy controls, the study seeks to determine whether FM patients show a higher prevalence of subclinical ventricular dysfunction.

The study is designed as a prospective, observational, case-control study. A total of 118 participants will be enrolled: 59 patients diagnosed with fibromyalgia according to the 2010 American College of Rheumatology (ACR) criteria, and 59 control subjects without fibromyalgia. The control group will consist of volunteers presenting with mechanical low back pain but without systemic rheumatic disease.

All participants will undergo echocardiographic examination using a standardized protocol with Vivid E95 Dimension ultrasound equipment (GE Healthcare). Global Longitudinal Strain will be measured offline using EchoPAC software, and results will be analyzed according to recommendations of the American Society of Echocardiography. In addition, fibromyalgia patients will complete the Fibromyalgia Impact Questionnaire (FIQ) to evaluate disease severity, and results will be compared with echocardiographic findings.

Primary Outcome: Prevalence of subclinical left ventricular dysfunction, defined as impaired GLS, in fibromyalgia patients compared to controls.

Secondary Outcome: Correlation between GLS values and fibromyalgia disease severity scores.

This study is expected to provide new insights into the cardiovascular involvement of fibromyalgia. Detecting early myocardial impairment with GLS may help identify patients at risk of future cardiovascular complications and may support closer monitoring and preventive strategies in this population.

DETAILED DESCRIPTION:
Fibromyalgia (FM) is a chronic, multisystem disorder affecting approximately 2-4% of the general population, predominantly women. It is characterized by widespread musculoskeletal pain, fatigue, sleep disturbances, anxiety, cognitive impairment, and autonomic symptoms such as gastrointestinal irregularities, Raynaud-like phenomena, and sicca complaints. The pathophysiology remains incompletely understood but is thought to involve central pain sensitization and dysautonomia.

Emerging evidence indicates that FM is associated with increased cardiovascular risk. Observational studies have demonstrated a higher prevalence of endothelial dysfunction, arterial stiffness, arrhythmias, and coronary artery disease in FM patients. Mechanistically, chronic sympathetic overactivity and persistent catecholamine release may increase myocardial oxygen demand, impair microvascular perfusion, and lead to subtle myocardial dysfunction. Autonomic imbalance has also been documented by heart rate variability studies, supporting impaired sympathetic-parasympathetic regulation. Importantly, the overlap between FM symptoms (fatigue, poor sleep, reduced functional capacity) and those of heart failure suggests a potential underrecognized cardiac component in FM.

Conventional echocardiography relies on left ventricular ejection fraction (LVEF) to evaluate systolic function. However, LVEF may remain normal despite underlying myocardial impairment and is strongly affected by loading conditions and observer variability. Many patients with heart failure present with preserved ejection fraction (HFpEF), underscoring the limitations of LVEF as an early marker of myocardial dysfunction.

Global Longitudinal Strain (GLS), assessed using two-dimensional speckle-tracking echocardiography (2D-STE), has emerged as a more sensitive and reproducible tool for detecting early myocardial dysfunction. GLS abnormalities can precede measurable reductions in LVEF and have prognostic value across diverse conditions including ischemic heart disease, hypertension, valvular disease, chemotherapy-related cardiotoxicity, and heart failure.

Preliminary studies in FM populations suggest possible subclinical myocardial involvement. Some reports describe increased risk of diastolic dysfunction and impaired GLS in FM patients, possibly reflecting the impact of chronic stress and autonomic dysregulation on cardiac mechanics. Nevertheless, systematic and adequately powered investigations remain scarce.

This prospective, observational, case-control study is designed to fill this knowledge gap. The study will enroll 59 FM patients diagnosed according to the 2010 American College of Rheumatology (ACR) criteria and 59 age- and sex-matched controls without systemic rheumatic disease. Echocardiographic examinations will be performed using a standardized protocol (Vivid E95, GE Healthcare), and GLS will be measured offline with EchoPAC software, following the American Society of Echocardiography guidelines. Disease severity in FM will be assessed using the Fibromyalgia Impact Questionnaire (FIQ).

The primary hypothesis is that FM patients will demonstrate a higher prevalence of impaired GLS, consistent with subclinical ventricular dysfunction, compared with controls. The secondary hypothesis is that higher FIQ scores will correlate with greater impairment in GLS, suggesting a relationship between disease burden and cardiac involvement.

The anticipated significance of this research lies in clarifying the cardiovascular component of fibromyalgia. Early identification of myocardial dysfunction using GLS may allow for improved risk stratification, closer clinical monitoring, and preventive strategies aimed at reducing long-term cardiovascular morbidity. Beyond its clinical relevance, this study also extends the application of GLS into a non-traditional, rheumatology-related context, reinforcing the systemic nature of FM and the need for interdisciplinary management approaches.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50 years.
* No diagnosis of fibromyalgia.
* Volunteers presenting with mechanical low back pain but otherwise healthy.

Exclusion Criteria:

* Hypertension.
* Coronary artery disease.
* Diabetes mellitus.
* Significant valvular heart disease.
* Documented arrhythmias.
* Congestive heart failure.
* Systemic rheumatic diseases (e.g., SLE, RA).
* Hyperthyroidism or hypothyroidism.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients aged 18-50 years diagnosed with fibromyalgia according to the 2010 ACR criteria recruited from the Physical Medicine and Rehabilitation outpatient clinic of Ankara Training and Research Hospital, and age- and sex-matched healthy controls presenting with mechanical low back pain but without systemic disease.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-02-16 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Global Longitudinal Strain (GLS) in Fibromyalgia Patients | At the time of echocardiographic examination (Day 1, single assessment).
  Evaluation of left ventricular myocardial function by measuring Global Longitudinal Strain (GLS) using two-dimensional speckle-tracking echocardiography. GLS values of fibromyalgia patients will be compared with those of healthy controls to assess the presence of subclinical ventricular dysfunction.

SECONDARY OUTCOMES:
Correlation Between Global Longitudinal Strain (GLS) and Fibromyalgia Impact Questionnaire (FIQ) Scores | At the time of clinical and echocardiographic assessment (Day 1).
  The relationship between GLS values and disease severity will be evaluated by correlating echocardiographic GLS with the Fibromyalgia Impact Questionnaire (FIQ). The FIQ ranges from 0 to 100, with higher scores indicating worse disease impact. It is hypothesized that higher FIQ scores will correlate with impaired GLS values (less negative strain).
Prevalence of Subclinical Ventricular Dysfunction in Fibromyalgia Patients | At the time of echocardiographic examination (Day 1).
  The proportion of fibromyalgia patients with impaired GLS (< -18%) compared to healthy controls will be calculated to estimate the prevalence of subclinical ventricular dysfunction in the study population.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Therapy and Rehabilitation, University of Health Sciences, Ankara Training and Research Hospital, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to institutional policies regarding patient privacy and data protection regulations

REFERENCES:
- [Background] Chang KV, Hung CH, Sun WZ, Wu WT, Lai CL, Han DS, Chen CC. Evaluating soreness symptoms of fibromyalgia: Establishment and validation of the Revised Fibromyalgia Impact Questionnaire with Integration of Soreness Assessment. J Formos Med Assoc. 2020 Jul;119(7):1211-1218. doi: 10.1016/j.jfma.2019.10.018. Epub 2019 Nov 9. PMID 31711726
- [Background] Galvez-Sanchez CM, Reyes Del Paso GA. Diagnostic Criteria for Fibromyalgia: Critical Review and Future Perspectives. J Clin Med. 2020 Apr 23;9(4):1219. doi: 10.3390/jcm9041219. PMID 32340369
- [Background] Rong LQ, Neuburger PJ, Kim J, Devereux RB. Left ventricular global longitudinal strain and cardiac surgical outcomes. Minerva Cardioangiol. 2020 Oct;68(5):489-496. doi: 10.23736/S0026-4725.20.05251-2. Epub 2020 May 29. PMID 32472988
- [Background] Tschope C, Senni M. Usefulness and clinical relevance of left ventricular global longitudinal systolic strain in patients with heart failure with preserved ejection fraction. Heart Fail Rev. 2020 Jan;25(1):67-73. doi: 10.1007/s10741-019-09853-7. PMID 31489515
- [Background] Ueyama H, Kuno T, Takagi H, Krishnamoorthy P, Prandi FR, Palazzuoli A, Sharma SK, Kini A, Lerakis S. Prognostic value of left ventricular global longitudinal strain in mitral regurgitation: a systematic review. Heart Fail Rev. 2023 Mar;28(2):465-483. doi: 10.1007/s10741-022-10265-3. Epub 2022 Jul 28. PMID 35900680
- [Background] Smiseth OA, Rider O, Cvijic M, Valkovic L, Remme EW, Voigt JU. Myocardial Strain Imaging: Theory, Current Practice, and the Future. JACC Cardiovasc Imaging. 2025 Mar;18(3):340-381. doi: 10.1016/j.jcmg.2024.07.011. Epub 2024 Sep 11. PMID 39269417
- [Background] Velagapudi VM, Pidikiti R, Tighe DA. Is Left Ventricular Global Longitudinal Strain by Two-Dimensional Speckle Tracking Echocardiography in Sepsis Cardiomyopathy Ready for Prime Time Use in the ICU? Healthcare (Basel). 2019 Jan 3;7(1):5. doi: 10.3390/healthcare7010005. PMID 30609787
- [Background] Potter E, Marwick TH. Assessment of Left Ventricular Function by Echocardiography: The Case for Routinely Adding Global Longitudinal Strain to Ejection Fraction. JACC Cardiovasc Imaging. 2018 Feb;11(2 Pt 1):260-274. doi: 10.1016/j.jcmg.2017.11.017. PMID 29413646
- [Background] Cho KI, Lee JH, Lee HG, Kim SM, Kim TI. Assessment of myocardial function in patients with fibromyalgia and the relationship to chronic emotional and physical stress. Korean Circ J. 2010 Feb;40(2):74-80. doi: 10.4070/kcj.2010.40.2.74. Epub 2010 Feb 23. PMID 20182592
- [Background] Sayilir S, Ergun G, Ekiz T. Evaluation of Ventricular Diastolic Function in Patients With Fibromyalgia Syndrome. Arch Rheumatol. 2017 Aug 15;33(2):150-153. doi: 10.5606/ArchRheumatol.2018.6541. eCollection 2018 Jun. PMID 30207569
- [Background] Gist AC, Guymer EK, Ajani AE, Littlejohn GO. Fibromyalgia has a high prevalence and impact in cardiac failure patients. Eur J Rheumatol. 2017 Dec;4(4):245-249. doi: 10.5152/eurjrheum.2017.17026. Epub 2017 Nov 2. PMID 29308277
- [Background] Zetterman T, Markkula R, Miettinen T, Kalso E. Heart rate variability responses to cognitive stress in fibromyalgia are characterised by inadequate autonomous system stress responses: a clinical trial. Sci Rep. 2023 Jan 13;13(1):700. doi: 10.1038/s41598-023-27581-9. PMID 36639565
- [Background] Su CH, Chen JH, Lan JL, Wang YC, Tseng CH, Hsu CY, Huang L. Increased Risk of Coronary Heart Disease in Patients with Primary Fibromyalgia and Those with Concomitant Comorbidity-A Taiwanese Population-Based Cohort Study. PLoS One. 2015 Sep 14;10(9):e0137137. doi: 10.1371/journal.pone.0137137. eCollection 2015. PMID 26366998
- [Background] Tsai PS, Fan YC, Huang CJ. Fibromyalgia is associated with coronary heart disease: a population-based cohort study. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):37-42. doi: 10.1097/AAP.0000000000000190. PMID 25436616
- [Background] Sethi P, Peiris CD. A Review of Catecholamine Associated Cardiomyopathies and Channelopathies. Cureus. 2020 Feb 11;12(2):e6957. doi: 10.7759/cureus.6957. PMID 32195067
- [Background] Kocyigit BF, Akyol A. Coexistence of fibromyalgia syndrome and inflammatory rheumatic diseases, and autonomic cardiovascular system involvement in fibromyalgia syndrome. Clin Rheumatol. 2023 Mar;42(3):645-652. doi: 10.1007/s10067-022-06385-8. Epub 2022 Sep 23. PMID 36151442
- [Background] Kulshreshtha P, Deepak KK, Yadav RK, Mukherjee D. Cardiac autonomic neuropathy in fibromyalgia: Revisited. J Back Musculoskelet Rehabil. 2022;35(1):111-117. doi: 10.3233/BMR-200209. PMID 34092594